CLINICAL TRIAL: NCT04403464
Title: The Effect of Using a New Interactive Device Based on Motor Skill Learning Principles on the Motor and Functional Abilities of Children With Bilateral Cerebral Palsy
Brief Title: Effect of a New Interactive Device on the Motor and Functional Abilities of Children With Bilateral Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B403201316810e
Record Dates: First submitted 2020-05-20; First posted 2020-05-27 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy
Keywords: motor skill learning; intensive therapy; selective voluntary motor control; cerebral palsy; assistive technology; therapeutic device
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT-ILE with REAtouch® (Experimental): Hand and Arm Bimanual Intensive Therapy Including Lower Extremities with an interactive device
  Interventions: Behavioral: HABIT-ILE with REAtouch®
- HABIT-ILE without REAtouch® (Active Comparator): Hand and Arm Bimanual Intensive Therapy Including Lower Extremities
  Interventions: Behavioral: HABIT-ILE without REAtouch®

INTERVENTIONS:
Behavioral: HABIT-ILE with REAtouch® — 65h HABIT-ILE including 30h REAtouch®
  Arms: HABIT-ILE with REAtouch®
Behavioral: HABIT-ILE without REAtouch® — 65h HABIT-ILE
  Arms: HABIT-ILE without REAtouch®

SUMMARY:
Recent research has shown that interventions with assistive technologies lead to an improvement in the motor and functional abilities of children with cerebral palsy (CP). REAtouch® is a new interactive interface based on motor skill learning principles. Its efficiency during intensive motor skill learning interventions has never been tested in children with bilateral cerebral palsy.

Therefore, the study aims to investigate the efficiency of using a virtual reality tool to provide a motor skill learning intervention in a randomized trial.

DETAILED DESCRIPTION:
Recent research has shown that interventions with assistive technologies could lead to an improvement in the motor and functional abilities of children with cerebral palsy (CP). However they usually miss the functional motor skill learning qualities to match the changes observed in high intensity motor skill learning based interventions.REAtouch® is a new interactive interface based on motor skill learning principles that could be implemented in intensive interventions.

Therefore, the study aims to investigate the effects of intensive interventions with or without the interface on the motor and functional abilities of children with bilateral CP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed bilateral cerebral palsy,
* MACS levels from I to III,
* GMFCS levels from I to III,
* Ability to follow instructions and complete testing.

Exclusion Criteria:

* Orthopedic surgery, botulinum toxin injections or another unusual intervention less than 6 months before or within the study period.
* Unstable seizure
* Severe visual or cognitive impairments likely to interfere with intervention or testing session completion

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in Gross Motor Function Measure (GMFM-66): | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The GMFM has been developed to measure the change in gross motor function over time in children with cerebral palsy.
Changes in ABILHAND-Kids Questionnaire | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  This ABILHAND-Kids Questionnaire has been developed to assess a child's unimanual and bimanual upper limb activities. It ranges from - 6 to +6 logits (higher score means better performance).

SECONDARY OUTCOMES:
Changes in Test of Arm Selective Control (TASC) | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The TASC is an upper limb selective motor control evaluation tool including eight motions in each arm and up to three attempts are allowed for each motion. After completion of the best attempt, points ranging from 0 (absent), 1 (impaired) to 2 (normal) are recorded for each joint depending on the movement properties and descriptors of the test.
Changes in Selective Control Assessment of the Lower Extremity (SCALE) | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The SCALE was designed to evaluate lower limb selective motor control of children with cerebral palsy. The SCALE includes testing of five reciprocal lower extremity movements. SVMC is graded at each joint as 'Normal' (2 points), 'Impaired' (1 point), or 'Unable' (0 points).
Changes in 6 Minutes Walking Test (6MWT) | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The 6 Minutes Walking Test measures the distance that the patient walk as much as possible within a period of 6-minutes in a 30 meters long corridor.
Changes in Box and Blocks test (BBT) | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The BBT is a test of gross manual dexterity. Each hand is tested individually and the BBT is scored through the number of blocks carried over the partition from one part to another part of a box during the one-minute trial period.
Changes in Jebsen-Taylor Test | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The Jebsen-Taylor Test assesses uni-manual hand function, through 7 subtests simulating daily life activities. The test assesses speed, not quality of performance and time to complete each activity is reported using a stopwatch.
Changes in Modified Cooper test | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The Modified Cooper test is a modified version of The Manual Form Perception Test, which evaluates stereognosis through 16 objects. Both hands are tested separately and time to recognise the objects is reported using a stopwatch.
Changes in ACTIVLIM-CP Questionnaire | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The ACTIVLIM-CP Questionnaire measures a patient's ability to perform daily activities requiring the use of the upper and/or the lower limbs through 42 items specific to patients with cerebral palsy. It ranges from - 5 to +5 logits (higher score means better performance).
Changes in ABILOCO-Kids Questionnaire | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The ABILOCO-Kids Questionnaire measures a patient's ability to perform daily activities requiring the use of the lower limbs through 10 items specific to patients with cerebral palsy. It ranges from - 4 to +4 logits (higher score means better performance).
Changes in Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The PEDI-CAT is the new version of the Pediatric Evaluation of Disability Inventory (PEDI). The PEDI-CAT is comprised of 276 functional activities acquired throughout infancy, childhood and young adulthood. Based on the nternational Classification of Functioning, Disability and Health for Children and Youth (ICF-CY) model, the PEDI-CAT contents provide information about the activities and participation component. It ranges from 0 to 100% (higher score means better performance).
Changes in Canadian Occupational Performance Measure (COPM) | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The COPM measures the patient's self-perception of occupational performance and satisfaction of it in daily activities over time. It ranges from 1 to 10 (higher score means better performance).
Changes in Both Hands Assessment (BoHA) | pre-camp (1 week before), post-camp (1 week after), 3 months follow- up
  The BoHA is a videotaped tool measuring how effectively children with bilateral CP use both hands in bimanual activities.
Changes in Executive Functions | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Cognitive functions of the children will be assessed by Stroop task and Flanker task.
Changes in spatial parameters of the gait (Kinematics assessments) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the stride length (meters), step length (meters) and step width (meters).
Changes in temporal parameters of the gait (Cycle time) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the cycle of gait time (seconds).
Changes in temporal parameters of the gait (Stance time) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the stance time (percentage of the total gait cycle).
Changes in temporal parameters of the gait (Swing time) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the swing time (percentage of the total gait cycle).
Changes in temporal parameters of the gait (Stride) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the gait cadence (stride per minute).
Changes in temporal parameters of the gait (Velocity) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the gait velocity (meter/second).
Changes in temporal parameters of the gait (Acceleration) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the gait acceleration (meters/second^2).
Changes in spatial parameters of the upper extremity (Straightness) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the straightness (percentage of upper extremity trajectory during a reaching task).
Changes in spatial parameters of the upper extremity (Smoothness) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the smoothness (variability of the movement during a reaching task)
Changes in temporal parameters of the upper extremity (Kinematics assessments) | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Through a 3D motion system, we measure the time from onset to end of the task (seconds). the task consists in a reaching task.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, Professor, Principal Investigator — Institute of Neuroscience, UCLouvain
Locations (1):
- Institute of Neuroscience, UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No